CLINICAL TRIAL: NCT03751995
Title: POEM (Practice of Embracing Each Moment) Study (Delivery Science)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CN-18-3183
Record Dates: First submitted 2018-08-23; First posted 2018-11-23 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Advanced Cancer; Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: pilot pragmatic cluster randomized trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants from medical centers assigned to the control arm will receive usual care.
- Intervention (Experimental): Participants from medical centers assigned to the intervention arm will receive access to their choice of a mindfulness app or a webinar-based mindfulness course for 6 weeks.
  Interventions: Behavioral: Mindfulness meditation

INTERVENTIONS:
Behavioral: Mindfulness meditation — Participants in the intervention group will have their choice of two commercially available mindfulness programs, HeadspaceTM and eMindful for 6 weeks.
  The Headspace program provides progressive guided mindfulness meditation instruction via a website and mobile app to help users learn the skills of mindfulness for use in everyday life. Sessions last 3-20 minutes. Videos encourage the integration of mindfulness into daily life.
  eMindful offers an online virtual classroom where participants can participate in synchronous, 1-hour mindfulness classes 1-2 times per week. The program is modeled after the mindfulness-based stress reduction (MBSR) program. eMindful also offers a cancer-specific meditation course that participants may choose to participate in.
  Arms: Intervention

SUMMARY:
The objective of the proposed pilot pragmatic cluster randomized trial targeting cancer patients undergoing palliative and supportive therapy and their informal caregivers is to pilot test implementation of mHealth two mindfulness interventions as part of standard palliative care support within Kaiser Permanente Northern California.

DETAILED DESCRIPTION:
A cancer diagnosis is associated with high levels of distress in both patients and their family caregivers. Although studies have demonstrated that mindfulness-based interventions are effective in reducing distress and anxiety of cancer patients, logistical limitations of currently available mindfulness-based stress reduction training options restrict their potential to benefit patients with advanced cancer and their caregivers. Previous pilot mindfulness studies targeting cancer patients and caregivers have demonstrated preliminary feasibility and acceptability of mHealth mindfulness interventions and preliminary efficacy in reducing depression, anxiety and improving quality of life. The objective of the proposed pilot pragmatic cluster randomized trial targeting cancer patients undergoing palliative and supportive therapy and their informal caregivers is to pilot test implementation of two mHealth mindfulness interventions as part of standard palliative care support within KPNC. Using data collected through the mindfulness programs, patient/caregiver surveys, clinician surveys, and EHR data, the study aims are: 1) to assess acceptability and feasibility of incorporating an mHealth mindfulness intervention as part of palliative care and to obtain preliminary efficacy of the intervention on patient-reported outcomes, clinical outcomes, and health care utilization; and 2) to gather qualitative feedback regarding the intervention from the clinicians, patients and caregivers. Participating oncology clinics will be randomized into either intervention or usual care arms. Intervention participants may choose from a 6-week webinar-based mindfulness program or a 6-week self-paced mobile app-based mindfulness program. Controls will receive usual care. Rates of participation, completion and adherence among intervention participants and participant-reported outcomes on distress and quality of life among both arms at baseline, post-intervention and 12 weeks will be collected. The hypothesis is that participants in the intervention arm will experience reductions in depression/anxiety and improvement in immune function and quality of life. Clinician surveys and interviews with intervention participants will also be conducted at the end of the intervention to obtain feedback regarding the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Smartphone or tablet ownership OR has a computer with internet access
* Ability to read and understand English
* Patients: current Kaiser Permanente member with diagnosis of cancer and receiving palliative or supportive therapy at one of the participating oncology clinics
* Caregivers: primary unpaid support person of the patient who takes care of the patient at least two hours a week.

Exclusion Criteria:

* Severe hearing impairment
* Severe mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2020-04-29 (Actual)

PRIMARY OUTCOMES:
Change in Hospital Anxiety and Depression Scale | Baseline to 6 weeks
  The 14-item Hospital Anxiety and Depression Scale (HADS) assesses anxiety and depression. Each subscale (depression and anxiety) is scored from 0 to 21 by summing individual item scores, with higher scores indicating greater anxiety and depression; 0-7 is generally considered within normal range.
Change in Hospital Anxiety and Depression Scale | Baseline to 12 weeks
  The 14-item Hospital Anxiety and Depression Scale (HADS) assesses anxiety and depression. Each subscale (depression and anxiety) is scored from 0 to 21 by summing individual item scores, with higher scores indicating greater anxiety and depression; 0-7 is generally considered within normal range.

SECONDARY OUTCOMES:
Change in Functional Assessment of Chronic Illness Therapy-Palliative care (patients only) | Baseline to 6 weeks
  The 46-item Functional Assessment of Chronic Illness Therapy-Palliative care questionnaire assesses health-related quality of life for patients receiving palliative care. It includes subscales for physical, social, emotional and functional well-being as well as a fifth subscale for additional item relevant to quality of life for persons with advanced or life-limiting illness. Scores are calculated by summing the scores from the individual items for the overall score or from the individual items in each subscale for the subscale scores. The score can range from 0 to 184 for the overall scale, 0-76 for the palliative care items, 0-28 for the physical, social, and functional well-being subscales, and 0-24 for the emotional well-being subscale. Higher scores indicate better quality of life.
Change in Functional Assessment of Chronic Illness Therapy-Palliative care (patients only) | Baseline to 12 weeks
  The 46-item Functional Assessment of Chronic Illness Therapy-Palliative care questionnaire assesses health-related quality of life for patients receiving palliative care. It includes subscales for physical, social, emotional and functional well-being as well as a fifth subscale for additional item relevant to quality of life for persons with advanced or life-limiting illness. Scores are calculated by summing the scores from the individual items for the overall score or from the individual items in each subscale for the subscale scores. The score can range from 0 to 184 for the overall scale, 0-76 for the palliative care items, 0-28 for the physical, social, and functional well-being subscales, and 0-24 for the emotional well-being subscale. Higher scores indicate better quality of life.
Change in Brief COPE coping strategy questionnaire (patients only) | Baseline to 6 weeks
  The Brief COPE is a 28-item questionnaire that measures coping strategies. There are 14 scales with 2 items each: self-distraction, active coping, denial, substance use, use of emotional support, use of instrumental support, behavioral disengagement, venting, positive reframing, planning, humor, acceptance, religion, and self-blame. Items are summed to produce scale scores (possible range: 2-8), with higher scores reflecting greater use of a particular coping strategy.
Change in Brief COPE coping strategy questionnaire (patients only) | Baseline to 12 weeks
  The Brief COPE is a 28-item questionnaire that measures coping strategies. There are 14 scales with 2 items each: self-distraction, active coping, denial, substance use, use of emotional support, use of instrumental support, behavioral disengagement, venting, positive reframing, planning, humor, acceptance, religion, and self-blame. Items are summed to produce scale scores (possible range: 2-8), with higher scores reflecting greater use of a particular coping strategy.
Change in Post-Traumatic Growth Inventory | Baseline to 6 weeks
  The 21-item Posttraumatic Growth Inventory (PTGI) assesses five factors of posttraumatic growth (positive change experienced because of a traumatic event or crisis): relating to others (7 items), new possibilities (5 items), personal strength (4 items), spiritual change (2 items), and appreciation of life (3 items). Respondents are asked to rate to what extent they have seen the listed changes as a result as a crisis in their lives. The PTGI is scored by adding all the responses (score range: 0-105). Individual factors are scored by adding responses to items on each factor (score range: 0-(number of items x 5)).
Change in Post-Traumatic Growth Inventory | Baseline to 12 weeks
  The 21-item Posttraumatic Growth Inventory (PTGI) assesses five factors of posttraumatic growth (positive change experienced because of a traumatic event or crisis): relating to others (7 items), new possibilities (5 items), personal strength (4 items), spiritual change (2 items), and appreciation of life (3 items). Respondents are asked to rate to what extent they have seen the listed changes as a result as a crisis in their lives. The PTGI is scored by adding all the responses (score range: 0-105). Individual factors are scored by adding responses to items on each factor (score range: 0-(number of items x 5)).
Change in Five Facet Mindfulness Questionnaire | Baseline to 6 weeks
  The 24-item Five Facet Mindfulness Questionnaire (short form) (FFMQ) measures five factors representing elements of mindfulness: observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. Factor subscale scores are calculated by summing individual items scores and range from 5-25 except for the 'observing' subscale, which ranges 4-20. Higher scores indicate greater mindfulness.
Change in Five Facet Mindfulness Questionnaire | Baseline to 12 weeks
  The 24-item Five Facet Mindfulness Questionnaire (short form) (FFMQ) measures five factors representing elements of mindfulness: observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. Factor subscale scores are calculated by summing individual items scores and range from 5-25 except for the 'observing' subscale, which ranges 4-20. Higher scores indicate greater mindfulness.
Change in Caregiver Quality of Life-Cancer scale (caregivers only) | Baseline to 6 weeks
  The Caregiver Quality of Life Index - Cancer (CQOLC) 35-item scale gauges the daily and overall impact caregiving has on respondents' quality of life. The overall score is calculated by summing all items, and possible scores range 0-140. Higher scores indicate better quality of life.
Change in Caregiver Quality of Life-Cancer scale (caregivers only) | Baseline to 12 weeks
  The Caregiver Quality of Life Index - Cancer (CQOLC) 35-item scale gauges the daily and overall impact caregiving has on respondents' quality of life. The overall score is calculated by summing all items, and possible scores range 0-140. Higher scores indicate better quality of life.
Change in PROMIS pain interference scale (caregivers only) | Baseline to 6 weeks
  The 9-item PROMIS Pain Interference scale assesses pain level and extent to which pain interfered with functional activities during the past 7 days. The pain base score is based on one item and scores range 0-10. The pain interference is calculated by summing the remaining 8 items and scores range 8-40.
Change in PROMIS pain interference scale (caregivers only) | Baseline to 12 weeks
  The 9-item PROMIS Pain Interference scale assesses pain level and extent to which pain interfered with functional activities during the past 7 days. The pain base score is based on one item and scores range 0-10. The pain interference is calculated by summing the remaining 8 items and scores range 8-40.
Change in PROMIS sleep disturbance scale (caregivers only) | Baseline to 6 weeks
  The 8-item PROMIS Sleep Disturbance scale assesses sleep disturbance during the past 7 days. A higher summary score, calculated by summing scores from individual items, indicates worse sleep disturbance. Possible scores range from 8-40.
Change in PROMIS sleep disturbance scale (caregivers only) | Baseline to 12 weeks
  The 8-item PROMIS Sleep Disturbance scale assesses sleep disturbance during the past 7 days. A higher summary score, calculated by summing scores from individual items, indicates worse sleep disturbance. Possible scores range from 8-40.
Change in Brief Fatigue Inventory (caregivers only) | Baseline to 6 weeks
  The 9-item Brief Fatigue Inventory (BFI) assesses the severity and impact of fatigue and the extent to which fatigue interfered with various aspects of life in the past 24 hours (e.g., mood) on a 10-point Likert scale. A global fatigue score can be obtained by averaging all the items on the BFI (score range: 0-10). Higher scores on the BFI correspond to greater self-reported levels of fatigue.
Change in Brief Fatigue Inventory (caregivers only) | Baseline to 12 weeks
  The 9-item Brief Fatigue Inventory (BFI) assesses the severity and impact of fatigue and the extent to which fatigue interfered with various aspects of life in the past 24 hours (e.g., mood) on a 10-point Likert scale. A global fatigue score can be obtained by averaging all the items on the BFI (score range: 0-10). Higher scores on the BFI correspond to greater self-reported levels of fatigue.
Change in Distress Thermometer | Baseline to 6 weeks
  The National Comprehensive Cancer Network Distress Thermometer assesses current distress level. Respondents are asked to rate their level of distress during the past week by choosing a number, with 0 indicating no distress and 10 extreme distress.
Change in Distress Thermometer | Baseline to 12 weeks
  The National Comprehensive Cancer Network Distress Thermometer assesses current distress level. Respondents are asked to rate their level of distress during the past week by choosing a number, with 0 indicating no distress and 10 extreme distress.

CONTACTS AND LOCATIONS:
Overall Officials: Ai Kubo, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Northern California, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No